CLINICAL TRIAL: NCT02656511
Title: Immediate Initiation of Antiretroviral Therapy During Acute HIV Infection
Brief Title: Immediate Initiation of Antiretroviral Therapy During "Hyperacute" HIV Infection
Acronym: DGVTAF
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: ViiV Healthcare (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-236-1354
Record Dates: First submitted 2015-12-31; First posted 2016-01-15 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: HIV
Keywords: immediate antiretroviral therapy; hyperacute infection
MeSH Terms: interventions — dolutegravir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dolutegravir+Emtricitabine/Tenofovir (Experimental): Dolutegravir 50 mg PO daily plus Emtricitabine 200 mg/Tenofovir alafenamide 25 mg
  Interventions: Drug: Dolutegravir; Drug: Emtricitabine/Tenofovir

INTERVENTIONS:
Drug: Dolutegravir — Dolutegravir 50 mg PO daily
  Other Names: Tivicay
Drug: Emtricitabine/Tenofovir — Emtricitabine 200 mg/Tenofovir alafenamide 25 mg PO daily
  Other Names: Truvada

SUMMARY:
The purpose of this study is to identify and provide immediate antiretroviral therapy to a cohort of HIV-infected individuals with very early HIV infection (estimated date of infection within the last 90 days). The primary aim of the study is to evaluate whether initiation of dolutegravir plus emtricitabine/tenofovir during acute/early HIV infection leads to protection of CD4+ T cells and other immune cells in the peripheral blood and lymphoid tissue from infection.

DETAILED DESCRIPTION:
Although ART decreases HIV-associated mortality, it does not appear to completely restore immune health, for reasons that remain unclear. In addition, while HIV prevention approaches have led to significant successes in decreasing the incidence of new HIV infection over the past few years, the epidemic continues to grow both locally and globally. While complete eradication may not currently be feasible, a "functional cure" in which patients are able to indefinitely maintain undetectable viral loads in the absence of therapy may be an attainable immediate goal. Studying patients with early HIV infection and immediate ART will provide a unique opportunity to investigate the pathophysiology of the earliest stages of HIV infection and may help identify the virologic/immunologic predictors of a functional cure.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Male or female, age ≥18 years
3. Acute HIV infection with a negative or indeterminate HIV-1 antibody test and plasma HIV-1 RNA > 40 cp/ml, OR clinical history consistent with new HIV infection in the last 90 days.
4. Antiretroviral therapy untreated or recently initiated (within 7 days)
5. Participant must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.
6. All participants must agree not to participate in a conception process (eg, active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization)..
7. When participating in sexual activity that could lead to pregnancy, female participants must agree to use a double barrier method of contraception for at least two weeks after discontinuation of study drug.

Exclusion Criteria:

1. Known severe kidney disease (CrCl < 60 ml/min via Cockcroft-Gault method)
2. Known severe hepatic impairment (Child-Pugh Class C)
3. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
4. Participants with anticipated need for Hepatitis C virus (HCV) therapy during study
5. Concurrent treatment with dofetilide, oxcarbazepine, phenytoin, phenobarbital, carbamazepine, St. John's wort, or metformin
6. Serious illness requiring systemic treatment and/or hospitalization in the preceding 90 days prior to study enrollment
7. Concurrent treatment with immunomodulatory drugs, or exposure to any immunomodulatory drugs in the preceding 90 days prior to study enrollment (e.g. IL-2, interferon-alpha, methotrexate, cancer chemotherapy)
8. Concurrent treatment with investigational drugs, or exposure to any investigational drugs in the preceding 90 days prior to study enrollment
9. Active drug or alcohol use or dependence that, in the opinion of the Principal Investigator, would interfere with adherence to study requirements
10. Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation
11. Pregnant or breastfeeding women.
12. For participants who agree to colorectal biopsy
13. Known blood coagulation disorder
14. Platelets < 50,000/mm^3
15. PTT > 2x upper limit of normal
16. INR > 1.3
17. Use of aspirin, NSAIDs, Plavix, Coumadin, or other blood thinners that cannot be stopped for clinical reasons for 5 days before and after each colorectal biopsy
18. Inflammatory colitis (e.g., Crohn's disease and/or ulcerative colitis) and/or any contraindications to sigmoidoscopy or colorectal biopsy such as peritonitis, active diverticulitis, or recent bowel surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of immediate Dolutegravir plus Emtricitabine/Tenofovir administered to acutely infected HIV patients. | 6 months
  The number of grade 2 or higher severity adverse events (AEs) or drug-related laboratory abnormalities that exceed a frequency of 5% over a 6 month study period.

SECONDARY OUTCOMES:
Change in HIV reservoir size (cell-associated total DNA) in peripheral blood | 5 years
  The change in HIV reservoir size (as measured by cell-associated total DNA levels in peripheral blood mononuclear cells) over a 6 month study period.
Change in HIV reservoir size (cell-associated integrated DNA) in peripheral blood | 5 years
  The change in HIV reservoir size (as measured by cell-associated integrated DNA levels in peripheral blood mononuclear cells) over a 6 month study period.
Change in HIV reservoir size (cell-associated unspliced RNA) in peripheral blood | 5 years
  The change in HIV reservoir size (as measured by cell-associated unspliced RNA levels in peripheral blood mononuclear cells) over a 6 month study period.

OTHER OUTCOMES:
Change in HIV reservoir size (cell-associated total DNA) in blood CD4+ subsets | 6 months
  The change in HIV reservoir size (as measured by cell-associated total DNA levels in peripheral blood CD4+ T cell subsets) over a 6 month study period.
Change in HIV reservoir size (cell-associated integrated DNA) in blood CD4+ subsets | 5 years
  The change in HIV reservoir size (as measured by cell-associated integrated DNA levels in peripheral blood CD4+ T cell subsets) over a 6 month study period.
Change in HIV reservoir size (cell-associated unspliced RNA) in blood CD4+ subsets | 6 months
  The change in HIV reservoir size (as measured by cell-associated unspliced RNA levels in peripheral blood CD4+ T cell subsets) over a 6 month study period.
Change in HIV reservoir size (cell-associated total DNA) in GALT CD4+ subsets | 6 months
  The change in HIV reservoir size (as measured by cell-associated total DNA levels in gut-associated lymphoid tissue [GALT] CD4+ T cell subsets) over a 6 month study period.
Change in HIV reservoir size (cell-associated integrated DNA) in GALT CD4+ subsets | 5 years
  The change in HIV reservoir size (as measured by cell-associated integrated DNA levels in gut-associated lymphoid tissue [GALT] CD4+ T cell subsets) over a 6 month study period.
Change in HIV reservoir size (cell-associated unspliced RNA) in GALT CD4+ subsets | 5 years
  The change in HIV reservoir size (as measured by cell-associated unspliced RNA levels in gut-associated lymphoid tissue [GALT] CD4+ T cell subsets) over a 6 month study period.

CONTACTS AND LOCATIONS:
Overall Officials: Sulggi Lee, MD PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whitehill GD, Joy J, Marino FE, Krause R, Mallick S, Courtney H, Park K, Carey J, Hoh R, Hartig H, Pae V, Sarvadhavabhatla S, Donaire S, Deeks SG, Lynch RM, Lee SA, Bar KJ. Autologous neutralizing antibody responses after antiretroviral therapy in acute and early HIV-1. J Clin Invest. 2024 Apr 23;134(11):e176673. doi: 10.1172/JCI176673. PMID 38652564